CLINICAL TRIAL: NCT03772821
Title: Development of a Predictive Score for Local Complications of Femoral Bifurcation Surgery: Prospective Multicenter Cohort Study
Brief Title: Development of a Predictive Score for Local Complications of Femoral Bifurcation Surgery
Acronym: PROFA
Status: Terminated | Type: Observational
Why Stopped: lack of inclusions
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: STEINMETZ 2018
Record Dates: First submitted 2018-12-04; First posted 2018-12-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Femoral Bifurcation Surgery
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Between D0 and D90: local and general complications, demographic, clinical, paraclinical and biological data
Other: Incision/scar measurement — Between D0 and D90

SUMMARY:
No prospective study has yet evaluated the factors influencing the complications of femoral bifurcation surgery in France. Daily practice of investigators suggests that conventional surgical treatment has had a higher rate of local complications in recent years for a variety of reasons that remain to be assessed (aging, overweight, chronic renal failure, diabetes, or other), but as of yet, investigators do not have proof of such an effect. The proposed study would follow a prospective, continuous, multicentre cohort of patients to describe the type, frequency and factors that contribute to local and general complications of surgery on the femoral bifurcation. This information is essential in the choice of the best revascularization technique for the femoral artery, which is frequently the site used for interventions in vascular conditions.

Surgeries will be performed in the normal manner. The research will be based on medical data collected during patient management. A measurement of the incision/scar will be taken once the procedure has been performed, either immediately after surgery or after a period of time, during post-operative consultation. Participation in this research will last 3 months from the day of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has not opposed participation in the study
* Age > 18 years old
* All patients with an open surgical approach to the common femoral artery and/or femoral bifurcation, uni or bilateral, with or without endovascular or open procedure

Exclusion Criteria:

* Patient with homolateral surgery of the femoral triangle which has not yet healed
* Person subject to court-ordered protection (curatorship, guardianship)
* Pregnant, parturient or breastfeeding woman
* Adult unable to consent
* Patient who refuses to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a surgical approach to the common femoral artery or femoral tripod
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Presence of at least one of the following local complications: dehiscence alone, dehiscence with infection, superficial infection, deep infection, other (lymphorrhea, hematoma, lymphocele) | Between Day 0 and Day 90

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Jean Minjoz, Besançon
  - CH Colmar, Colmar
  - CHU Dijon Bourgogne, Dijon
  - CH Mâcon, Mâcon
  - GHR Mulhouse, Mulhouse
  - CHU Nancy, Nancy
  - CH Troyes, Troyes